CLINICAL TRIAL: NCT00928811
Title: One-year Exploratory Study to Evaluate the Safety of Partial Replacement of CNI With Chronic Administration of Simulect in de Novo Normal-risk Kidney Transplant Recipients Treated With MPA
Brief Title: Study to Evaluate the Safety of Chronic Administration of Simulect to Subjects Receiving a First Kidney Transplant
Acronym: Simulect
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Investigator left University 04/2010
Sponsor: Drexel University College of Medicine (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, cynthia gifford, Research Administrator, Drexel University
Organization: Drexel University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17718; CHI 621A (Other: Drexel)
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: End Stage Renal Disease
Keywords: Simulect; de novo kidney transplant subjects; calcineurin inhibitors; Prograf
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Other): Standard of care administration with Simulect (basiliximab)being administered as per induction therapy on day of transplant and day 4.
  Interventions: Drug: basiliximab
- Simulect (Experimental): Simulect (basiliximab) intravenously day of transplant and day 4.
  Chronic Simulect (basiliximab) administration monthly for one year duration.
  Concomitant decrease in Prograf administration.
  Interventions: Drug: basiliximab

INTERVENTIONS:
Drug: basiliximab — Simulect 20 mg intravenously day of transplant and day 4
  Other Names: Simulect
  Arms: Control
Drug: basiliximab — Simulect (basiliximab) 20mg intravenously day of transplant and day 4 post operatively. Then Monthly administration of Simulect (basiliximab) 40 mg intravenously for one year duration.
  Other Names: Simulect (basiliximab)
  Arms: Simulect

SUMMARY:
The study is undertaken to explore the safety of using Simulect at monthly dose intervals to reduce the need of high dose/level CNI's such as Prograf.

DETAILED DESCRIPTION:
The use of CNI's after kidney transplantation is associated with typical adverse effects such as potential contribution to progressive impairment of renal function, hypertension, and metabolic abnormalities. The study consists of a run-in phase (1 month),and treatment phase (11 months) and safety assessment phase (1 month).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-75
* First kidney transplant from a living or deceased donor
* Receiving CNI and MPA
* Able to tolerate full dose MPA
* Calculated glomerular filtration rate >=30ml/min by Cockcroft-Gault equation
* Able to tolerate renal graft biopsies
* Provided written, informed consent
* Females of childbearing potential must have a negative pregnancy test within 48 hours prior to the first Simulect administration

Exclusion Criteria:

* Known hypersensitivity to Simulect
* Current preformed PRA>10%
* Multi organ or second kidney transplant
* Use of any investigational immunosuppressive drug within 1 month of inclusion
* Female patients who are pregnant, lactating or of child bearing potential and not practicing two approved methods of birth control
* Known malignancy or history of malignancy other than excised basal or squamous cell carcinoma of the skin
* HBV, HCV, or HIV positive patients
* Current severe infection
* Receiving an organ from an extended criteria donor per United Network for Organ Sharing (UNOS) guidelines
* Dialysis dependent one month post transplant
* Live too far away from the transplant center for adequate follow up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the risk of sensitization against the chimeric antibody, Simulect. | one year

SECONDARY OUTCOMES:
To describe the pharmacokinetics of Simulect over the study course. | one year
To determine the absolute and relative number of CD25 receptors on T cells at the end of each dosing interval. | one year
To assess the difference in calculated and measured GFR. | one year
To assess the difference in biopsy proven acute rejection rates and the acute and chronic parameters (chronic allograft injury) on surveillance biopsies. | one year
To assess the difference in vital signs and lab abnormalities | one year
To determine the difference in incidence and severity of albuminuria/proteinuria | one year
To collect safety data on infections and malignancies | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mysore Anil S. Kumar, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Drexel University College of Medicine, Philadelphia, Pennsylvania, United States